CLINICAL TRIAL: NCT06944600
Title: The Role of Sleep Disorders in the Motoric and Cognitive Trajectories of Older Physically Frail Sarcopenic and Healthy Active Subjects
Brief Title: Impact of Sleep Disorders and Digital Support on Older People's Health
Acronym: SOMNUS-DARE
Status: Not yet recruiting | Type: Observational
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Marcello Giuseppe Maggio, MD, PhD, Full Professor in Internal and Geriatric Medicine, University of Parma
Other Study IDs: 262/2024/SPER/UNIPR
Record Dates: First submitted 2025-04-17; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Sleep Disorders; Frailty; Cognitive Impairment; Quality of Life; Ageing; Digital Health; Multidisciplinary Approach
MeSH Terms: conditions — Sleep Wake Disorders; Frailty; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Physically frail sarcopenic older subjects
- Healthy active older subjects

SUMMARY:
The goal of this observational study is to learn about the effects of sleep disorders on health and ageing in older people over the age of 65.

The main question it aims to answer is: How do sleep disorders impact the motoric and cognitive ageing trajectories of older individuals? Participants will undergo a set of instrumental, laboratory and clinical diagnostic examinations to comprehensively assess the impact of sleep disorders on health.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years;
* MMSE score adjusted by age and education ≥ 25/30;
* Absence of mobility-disability;
* Absence of need for assistance with Basic Activities of Daily Living (according to the ICFSR International Clinical Practice Guidelines).

Exclusion Criteria:

* Individuals with specific clinical conditions that make the intervention unsafe (I.e., severe diseases, unstable health status);
* Individuals whose adherence to the protocol might be low due to clinical (E.g., cognitive impairment, dialysis) and non-clinical (E.g., plans to relocate out of the study area within the next 3 years) reasons;
* Individuals unable or unwilling to provide informed consent;
* Consumption of more than 14 alcoholic drinks per week [one alcoholic drink (equal to 14.0 grams of pure alcohol) corresponds to 36 cc of beer (5% alcohol content), 24 cc of malt liquor (7% alcohol content), 15 cc of wine (12% alcohol content), 4.5 cc of distilled spirit or liquor (40% alcohol content)];
* Difficulty in communicating with the study staff due to speech, language, or (non-corrected) hearing and vision problems;
* Severe arthritis (E.g., awaiting joint replacement) that would interfere with the ability to fully participate in the study;
* Lung disease requiring regular use of supplemental oxygen;
* Severe cardiovascular disease (including New York Heart Association [NYHA] class III or IV, clinically significant congestive heart failure and valvular disease, history of cardiac arrest, presence of an implantable defibrillator or pacemaker, uncontrolled angina);
* Upper and/or lower extremity amputation;
* Peripheral arterial disease Lériche-Fontaine 3 or 4;
* Renal disease requiring dialysis;
* Current enrolment in another study involving lifestyle, nutrition, or pharmaceutical interventions;
* Further medical, psychiatric, or behavioural factors that in the judgment of the principal investigator may interfere with the study participation;
* Further possible illnesses affecting the life expectancy and reducing it to less than 24 months, corresponding to the study's length;
* Clinical judgment concerning safety or non-compliance, as well as the conditions for which the use of the Sleep Profiler is not recommended (sensitivity of skin or scalp and/or open wounds on the forehead or scalp, allergic reactions to extended exposure to synthetic fabrics (e.g., polyester, rayon), upper respiratory infection or congestion, head circumference less than 21 or greater than 25 inches, forehead vertical measurement (from top of eyebrows to hairline) less than or equal to 2 inches or horizontal measurement (from hairline to hairline) less than or equal to 6 inches).
* SPPB score <3 at baseline.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Physically frail sarcopenic and healthy active subjects, from 65 years of age, admitted to the geriatric and sleep medicine outpatient clinic, not demented and independent in the Basic Activities of Daily Living.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of physical and functional worsening | 12 months

SECONDARY OUTCOMES:
Prevalence and incidence of sarcopenia | 24 months
Prevalence of mild cognitive impairment (MCI) and cognitive frailty | 24 months
Incidence of mild cognitive impairment (MCI) and cognitive frailty | 24 months
Incidence of dementia in cognitive frail older individuals | 24 months
Prevalence and incidence of recognised pre-frailty conditions | 24 months
Prevalence and incidence of malnutrition, polypharmacy and multimorbidity | 24 months